CLINICAL TRIAL: NCT06675695
Title: Emulation of the FLAURA (NCT02296125) Trial Using Specialty Oncology Electronic Health Records Databases
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor, Brigham and Women's Hospital
Other Study IDs: 2022P002556-ENC-FLAURA
Record Dates: First submitted 2024-11-01; First posted 2024-11-05 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2024-11

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- New use of osimertinib: Exposure group
  Interventions: Drug: New use of osimertinib
- New use of erlotinib or gefitinib: Reference group
  Interventions: Drug: New use of erlotinib or gefitinib

INTERVENTIONS:
Drug: New use of osimertinib — New use of osimertinib described in electronic health records is used as the exposure.
  Groups: New use of osimertinib
Drug: New use of erlotinib or gefitinib — New use of "standard of care" described in electronic health records (erlotinib or gefitinib) dispensing claim is used as the reference.
  Groups: New use of erlotinib or gefitinib

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale emulation of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
Randomized controlled trials (RCTs) are generally regarded as the gold-standard of evidence for establishing efficacy of medical products. However, real-world data (RWD) are increasingly used to complement evidence coming from RCTs. Yet, to have confidence in the accuracy of RWD studies of oncology products and their outcomes, investigators need to know which questions can be validly answered, with which non-interventional study designs and analysis methods, given the data that is available. Building on a process based on the RCT DUPLICATE initiative, the trial emulation discussed in this protocol is part of the expansion project EmulatioN of Comparative Oncology trials with Real-world Evidence (ENCORE) which is specific to oncology and aims to emulate 12 randomized oncology RCTs using multiple EHR data sources.

The purpose of this protocol is to describe the emulation of the FLAURA trial in a study conducted using specialty oncology electronic health record data. FLAURA was a Phase III, double-blind, randomised study assessing the efficacy and safety of AZD9291 (= osimertinib, 80 mg orally, once daily) versus a standard of care (SoC) Epidermal Growth Factor Receptor (EGFR) Tyrosine Kinase Inhibitor (TKI) (either gefitinib [250 mg orally, once daily] or erlotinib [150 mg orally, once daily]) in patients with locally advanced or metastatic EGFR sensitizing mutation (EGFRm+) Non-small Cell Lung Cancer (NSCLC) who are treatment-naïve and eligible for first-line treatment with an EGFR-TKI.

The database study designed to emulate FLAURA trial will be a new-user active comparative study, where we will compare the effect of osimertinib versus SoC on overall survival among patients with locally advanced or metastatic EGFRm+ NSCLC who are treatment-naïve and eligible for first-line treatment with an EGFR-TKI.

This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) extension project ENCORE, being conducted at the Brigham and Women's Hospital, Harvard Medical School. It is intended to emulate, as closely as is possible in specialty oncology electronic health records data, the trial listed below/above. Although many features of the trial cannot be directly emulated using secondary healthcare data, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not emulable in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare data for emulation for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Market availability of osimertinib began April 18, 2018.

Study Period:

ENCORE database 1 (EDB1): Patient identification period: 01/01/2011-04/30/2024 with follow-up information through data cut-off date on 04/30/2024

ENCORE database 2 (EDB2): Follow-up information through 02/24/2023 (there is no specific time period restrictions for patient eligibility)

ENCORE database 4 (EDB4): Patient identification period: 10/01/2018-09/30/2023 with follow-up information through data cut-off date on 09/30/2023.

Inclusion Criteria:

* Age >= 18
* New users of first-line antineoplastic system therapy: osimertinib, gefitinib, or erlotinib for advanced/metastatic disease
* Mention of 'adenocarcinoma' histology ('non-squamous' in EDB1)
* Line of therapy setting needs to be 'advanced' (EDB1), 'metastatic' (EDB2) or there needs to be evidence of metastatic disease at time of treatment initiation (EDB4)
* Evidence of any EGFR mutation in the 180 days before/on treatment initiation
* Treatment needs to be first-line for advanced (EDB1) or metastatic (EDB2) disease or patients with prior exposure to any potential antineoplastic treatment commonly used in the advanced/metastatic NSCLC setting are excluded (EDB4)
* ECOG 0 or 1 in the 90 days before/on treatment initiation

Exclusion Criteria:

* Missing age
* Concurrent primary malignancies (EDB2)
* Missing date of diagnosis or clinician note in the EHR (EDB2)
* Only one visit at provider site (EDB2)
* Metastatic (includes leukemias and multiple myeloma) for a malignancy diagnosed prior to the malignancy of interest with the presence of low grade (inclusive of grades 1 and 2) neuroendocrine histology (EDB2)
* Participation in any clinical trial at any point in treatment history (EDB4)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced or metastatic EGFR sensitizing mutation (EGFRm+) Non-small Cell Lung Cancer (NSCLC) who are treatment-naïve and eligible for first-line treatment with an EGFR-TKI
Sampling Method: Non-Probability Sample
Enrollment: 4864 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Time to all-cause mortality (overall survival) | Through the earliest of outcome, censoring, or end of data (April 2024)
  Hazard ratio (95% CI)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Data from specialty oncology electronic health records database will be licensed and used under data use agreements that prohibit sharing of data or data derivatives.

DOCUMENTS (1):
  • Study Protocol (2024-10-30): https://cdn.clinicaltrials.gov/large-docs/95/NCT06675695/Prot_000.pdf